CLINICAL TRIAL: NCT03844035
Title: Clinical and Biochemical Evaluation of Oral Irrigation in Patients With Periimplant Mucositis
Brief Title: Impacts of Oral Irrigation in Patients With Periimplant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Burcu Ozkan Cetinkaya, Professor in Periodontology, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/1034
Record Dates: First submitted 2019-02-06; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Peri-implant Mucositis
Keywords: periimplant mucositis

STUDY DESIGN:
Intervention Model Description: Forty-five patients with periimplant mucositis having at least one implant (age range:45-60) were included in study. Study was planned as randomized, single-blind, parallel-design. Patients were divided into 3 equal groups; i)toothbrush+oral irrigator ii)toothbrush+interdental brush, iii)only toothbrush. After baseline examinations [Silness-Löe plaque index(PI), Löe-Silness gingival index(GI), probing pocket depth(PPD), clinical attachment level(CAL), bleeding on probing(BOP)], initial periodontal therapy was completed using full-mouth disinfection method. Periimplant crevicular fluid(PCF) were taken from patents to assess levels of interleukin-1beta(IL-1β), Transforming growth factor-beta(TGF- β), tissue-type plasminogen activator(t-PA), plasminogen activator inhibitor-1(PAI-1). Clinical records were repeated at 2, 4 and 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral irrigator group (Experimental): Fifteen patients using toothbrush and oral irrigator(oxytet oral irrigatör).All patients were told to use Modified Bass method of tooth brushing technique. PI, GI, PPD and CAL values were measured with William's probe (Hu-Fried, Chicago, IL, A.B.D) around the teeth and with plastic probe around the implants. All clinical parameters were evaluated on each of the six regions of the implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual).PICF was collected one day after the clinical examination from buccal aspects of the mesial and distal surfaces at the interproximal sites.Following the initial clinical records, all patients were performed full mouth instrumentation and described oral hygiene procedure according to their groups.
  Interventions: Diagnostic Test: Periimplant crevicular fluid (PICF) collection
- Interdental brush group (Experimental): Fifteen patients using toothbrush and interdental brush.All patients were told to use Modified Bass method of tooth brushing technique. PI, GI, PPD and CAL values were measured with William's probe (Hu-Fried, Chicago, IL, A.B.D) around the teeth and with plastic probe around the implants. All clinical parameters were evaluated on each of the six regions of the implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). PICF was collected one day after the clinical examination from buccal aspects of the mesial and distal surfaces at the interproximal sites. Following the initial clinical records, all patients were performed full mouth instrumentation and described oral hygiene procedure according to their groups.
  Interventions: Diagnostic Test: Periimplant crevicular fluid (PICF) collection
- Control group (Active Comparator): Fifteen patients using only toothbrush.All patients were told to use Modified Bass method of tooth brushing technique. PI, GI, PPD and CAL values were measured with William's probe (Hu-Fried, Chicago, IL, A.B.D) around the teeth and with plastic probe around the implants. All clinical parameters were evaluated on each of the six regions of the implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual). PICF was collected one day after the clinical examination from buccal aspects of the mesial and distal surfaces at the interproximal sites. Following the initial clinical records, all patients were performed full mouth instrumentation and described oral hygiene procedure according to their groups.
  Interventions: Diagnostic Test: Periimplant crevicular fluid (PICF) collection

INTERVENTIONS:
Diagnostic Test: Periimplant crevicular fluid (PICF) collection — Prior to PICF sampling, supragingival plaque was removed by sterile curets and, after air drying, the surfaces were isolated by cotton rolls. Filter paper strips (periopaper, proflow Inc., Amityville, New York, USA) were placed in sulcus for 30s. Care was taken not to avoid mechanical trauma and strips contaminated with blood or saliva were discarded. The absorbed PICF volume was estimated by a calibrated instrument (periotron 8000, proflow Inc., Amityville, NY, USA). Then, the strips were sealed into sterile tubes before freezing at -80⁰C. The readings were converted to an actual volume (µl) by reference to the standard curve.

SUMMARY:
The present study aimed to investigate clinically the cleaning effectiveness of different treatment modalities, that is, oral irrigator or interdental brush usage addition to routine brushing and examine TGF-β1, IL-1β, t-PA, and PAI-1 levels in periimplant crevicular fluid of patients with periimplant mucositis. The null hypothesis was that oral irrigators would be effective compared to interdental brush in the oral care of individuals who use implant-supported protheses.

DETAILED DESCRIPTION:
Detailed Description: Our aim was to evaluate efficacy of a manual tooth-brush with either interdental brush or oral irrigator in treatment of periimplant mucositis.

Material and Method: Forty-five patients with periimplant mucositis having at least one implant (age range:45-60) were included in study. Study was planned as randomized, single-blind, parallel-design. Patients were divided into 3 equal groups; i)toothbrush+oral irrigator ii)toothbrush+interdental brush, iii)only toothbrush. After baseline examinations [Silness-Löe plaque index(PI), Löe-Silness gingival index(GI), probing pocket depth(PPD), clinical attachment level(CAL), bleeding on probing(BOP)], initial periodontal therapy was completed using full-mouth disinfection method. Periimplant crevicular fluid(PCF) were taken from patents to assess levels of interleukin-1beta(IL-1β), Transforming growth factor-beta(TGF- β), tissue-type plasminogen activator(t-PA), plasminogen activator inhibitor-1(PAI-1). Clinical records were repeated at 2, 4 and 12 weeks.

The hypothesis of our study is that oral irrigators may be effective in oral care of individuals using an implant-supported prosthesis because of the ease of use.

ELIGIBILITY:
Inclusion Criteria:

* subject with no systemic diseases that affect oral tissues and the nature of plaque,
* with no professional cleaning for at least six months prior to baseline examination,
* with one or more implants (Straumann, Waldenburg, Switzerland) functioning at least 24 months before the start of the study
* having implants with BOP in at least two of the six regions
* The people who agreed to refrain from the use of any nonstudy dental device or oral care product for the study duration were included in the study

Exclusion Criteria:

Exclusion criteria

* subjects not cooperative,
* having disease associated with bacteremia,
* taking medication influencing gingival health (eg. dilantin, calcium channel blockers, cyclosporine, anticoagulants),
* using long-term antibiotic and anti-inflammatory agents,
* smokers and
* women who were pregnant and in lactation period

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-06-05 (Actual)

PRIMARY OUTCOMES:
Periimplant crevicular fluid level of IL-1β as a marker of gingival inflammation | through study completion, an average of 1 year
  Elevated levels of IL-1β in periimplant crevicular fluid have been associated with the destructive changes that occur in the inflamed human gingiva
Periimplant crevicular fluid level of TGF-β1 as a marker both of inflammatory phase and proliferative phase | through study completion, an average of 1 year
  TGF-β1 plays a role in the development and progression of periodontal diseases.
Periimplant crevicular fluid level of t-PA as a marker for clinical evaluation and efficacy of periodontal treatment | through study completion, an average of 1 year
  Higher levels of t-PA in periimplant crevicular fluid have been associated with gingivitis and periodontitis.
Periimplant crevicular fluid level of PAI-1 as a marker for clinical evaluation and efficacy of periodontal treatment | through study completion, an average of 1 year
  Higher levels of PAI-1 may be associated with progression of periodontitis

CONTACTS AND LOCATIONS:
Overall Officials: Burcu OZKAN CETINKAYA, Prof, Study Director — Ondokuzmayis University, Faculty of Dentistry, Department of Periodontology,; Sema TUTUNCUOGLU, Dr, Principal Investigator — Samsun Oral and Dental Health Hospital, Samsun, Turkey; Ferda PAMUK, Assoc. Prof., Study Chair — Beykent University, Faculty of Dentistry, Department of Periodontology; Bahattin AVCI, Assoc. Prof., Study Chair — Ondokuzmayis University, Faculty of Medicine Department of Biochemistry; Gonca Cayir KELES, Prof, Study Chair — Okan University, Faculty of Dentistry, Department of Periodontology; Muge LUTFIOGLU, Assoc. Prof., Study Chair — Ondokuzmayis University, Faculty of Dentistry, Department of Periodontology; Şevki GULER, Assist.Prof., Study Chair — Izzet Baysal University, Faculty of Dentistry, Department of Periodontology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tutuncuoglu S, Cetinkaya BO, Pamuk F, Avci B, Keles GC, Kurt-Bayrakdar S, Lutfioglu M. Clinical and biochemical evaluation of oral irrigation in patients with peri-implant mucositis: a randomized clinical trial. Clin Oral Investig. 2022 Jan;26(1):659-671. doi: 10.1007/s00784-021-04044-x. Epub 2021 Jul 12. PMID 34251534